CLINICAL TRIAL: NCT03792919
Title: Virological Response After Cessation of Long Term Anti-HBV Nucleos(t)Ide Analogues (NAs) vs. Keeping on NAs Among Chronic Hepatitis B (CHB) Patients
Brief Title: Cessation of Long Term NAs vs. Keeping on NAs Among CHB Patients (CNAVK)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VENI-1
Record Dates: First submitted 2019-01-01; First posted 2019-01-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 2 groups. Group 1: Stop current anti-HBV neucleos(t)ides treatment, Group 2: Keep on current anti-HBV nucleus(t)ides treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cessation of NAs treatment (Experimental): Chronic hepatitis B patients who meet the criteria to stop the current anti-HBV Neucleos(t)ides treatment will stop their NAs at the baseline of the clinical trial.
  Interventions: Drug: Stop current treatment (anti-HBV neucleos(t)ides)
- Keep on current NAs treatment (Active Comparator): Chronic hepatitis B patients who meet the criteria to stop anti-HBV Neucleos(t)ides treatment will choose to keep on their current NAs treatment from the baseline of the clinical trial.
  Interventions: Drug: Keep current treatment (anti-HBV neucleos(t)ides)

INTERVENTIONS:
Drug: Stop current treatment (anti-HBV neucleos(t)ides) — Stop the current anti-HBV neucleos(t)ides treatment among the CHB patients who meet the criteria the stopping rule of long term treatment.
  Arms: Cessation of NAs treatment
Drug: Keep current treatment (anti-HBV neucleos(t)ides) — Keep the current anti-HBV neucleos(t)ides treatment among the CHB patients who meet the criteria the stopping rule of long term treatment.
  Arms: Keep on current NAs treatment

SUMMARY:
To Identify the collected cases who can stop NAs safely with satisfactory clinical outcome including sustain viral remission and HBsAg clearance among chronic hepatitis B(CHB) patients.

DETAILED DESCRIPTION:
Nucleos(t)ides analogues(NAs) is a safe and effective treatment among chronic hepatitis B(CHB) patients with excellent tolerance. Entecavir or tenofovir mono therapy has been shown to achieve inhibition of HBV replication in almost all adherent patients. However, HBsAg loss rate is low even after long-term NAs treatment. Recent studies indicated that cessation of NAs treatment could increase HBsAg clearance rate. Identifying the collected cases who can stop NAs safely with satisfactory clinical outcome including sustain viral remission and HBsAg clearance is very important.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg positive, HBeAg negative, antibody to HBeAg-positive;
2. Stable administration of anti-HBV neucleos(t)ides analogue mono therapy for at least more than one and a half year;
3. Demonstration of undetectable HBV DNA on three occasions, each at least 6 months apart, which is consistent with the APASL stopping rule;
4. Patients read, understand the consent form, and signed the study consent.

Exclusion Criteria:

1. Patient with other liver diseases;
2. Patient with concurrent hepatitis viruses or HIV infection;
3. Patients are reluctant to stop their anti-HBV treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HBsAg clearance | From baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of HBsAg clearance during the off-treatment period

SECONDARY OUTCOMES:
Incidence of HBsAg seroconversion | From baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of HBsAg seroconversion during the off-treatment period
Incidence of sustain HBV viral submission | rom baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of sustain HBV viral submission during the off-treatment period
Incidence of sustain biological response | rom baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of sustain biological response during the off-treatment period
Incidence of hepatocellular carcinoma | rom baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of hepatocellular carcinoma during the off-treatment period
Incidence of Liver failure | rom baseline to the end of the fifth year after cessation of anti-HBV treatment.
  The incidence of Liver failure during the off-treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity & Health Research Centre, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No